CLINICAL TRIAL: NCT03396965
Title: The Efficacy of Mini-c-arm Fluoroscopy for the Closed Reduction of Distal Radius Fractures in Adults
Brief Title: Mini-C-Arm for Distal Radius Fractures in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Steven Dailey, Principal Investigator, University of Cincinnati
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2014-6554
Record Dates: First submitted 2018-01-05; First posted 2018-01-11 (Actual); Last update posted 2018-01-16 (Actual); Status verified 2018-01

CONDITIONS: Distal Radius Fracture
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Intervention Model Description: Patients randomized to fluoroscopically-aided reduction of fracture, versus no fluoroscopic guidance
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mini-c-arm (Experimental): Fluoroscopically aided reductions
  Interventions: Other: Mini-c-arm
- Standard (No Intervention)

INTERVENTIONS:
Other: Mini-c-arm — Fluoroscopy used to aid reduction of distal radius fracture
  Arms: Mini-c-arm

SUMMARY:
Determine efficacy of the use of mini-c-arm fluoroscopy for the closed reduction of isolated distal radius fractures in adult patients in the emergency department setting.

ELIGIBILITY:
Inclusion Criteria:

* Closed distal radius fracture requiring reduction

Exclusion Criteria:

* Open, other ipsilateral upper extremity fractures, pregnant, incarcerated, less than 18 yo

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2015-05; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Reduction quality | Immediately post reduction
  Fracture alignment measured on post-reduction radiographs

IPD SHARING:
Plan to Share IPD: No